CLINICAL TRIAL: NCT03352349
Title: Effect of Terlipressinum on the Portal Vein Pressure of Patients With Liver Tumor After Liver Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Terlipressinum PVP
Record Dates: First submitted 2017-11-18; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Portal Vein Pressure
Keywords: Terlipressinum; Portal Vein Pressure; Liver Tumor Resection
MeSH Terms: interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Terlipressinum (Experimental): If the PVP is over 12 mmHg after hepatectomy, 1mg of Terlipressinum was given to patients intravenously. If the portal vein pressure is decreased by 1 mmHg, then 2mg of Terlipressinum was continuously given every day in the next 4 days after liver resection.
  Interventions: Drug: Terlipressinum

INTERVENTIONS:
Drug: Terlipressinum — If the PVP is over 12 mmHg after hepatectomy, 1mg of Terlipressinum was given to patients intravenously. If the portal vein pressure is decreased by 1 mmHg, then 2mg of Terlipressinum was continuously given every day in the next 4 days after liver resection.

SUMMARY:
In this study, investigators aim to screen out the patients with portal hypertension by monitoring intraoperative PVP, and to decide the effect of Terlipressinum on the portal pressure after liver resection.

DETAILED DESCRIPTION:
Liver resection is a common treatment for liver tumors. But the incidence of postoperative liver failure after hepatectomy is as high as 9-18.6%, which results in relatively high mortality rate . Portal hypertension is considered as a contraindication for hepatectomy according to the guidelines of the European Society of Hepatology and the American Society of Hepatology. Recent studies found that patients with portal hypertension were more likely to have persistent liver failure and shorter long-term survival after liver resection operation, compared to patients without portal hypertension.

Most of liver cancer patients in China have disease backgroud including chronic hepatitis and cirrhosis. Among liver cancer patients, of which function is Child A or B and have indication for liver resection, 25% of them have portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receives liver resection.
2. PVP is more than 12mmHg in 5 minutes after liver resection.

Exclusion Criteria:

1. Age: <18, >75;
2. Portal vein tumor thrombus is confirmed by preoperative assays;
3. Obstruction of biliary tract;
4. Active hepatitis;
5. Previous history of myocardial infarction;
6. Previous history of chronic kidney disease;
7. Severe arrhythmia;
8. Any other contraindications of the Terlipressinum.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Portal vein pressure | 8 months
  The change of the portal vein pressure before and after the use of Terlipressinum.

SECONDARY OUTCOMES:
Incidence of hepatic dysfunction after hepatectomy | 8 months
Incidence of acute renal dysfunction after hepatectomy | 8 months
Adverse effect of Terlipressurinum | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD&PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Background] Chen X, Zhai J, Cai X, Zhang Y, Wei L, Shi L, Wu D, Shen F, Lau WY, Wu M. Severity of portal hypertension and prediction of postoperative liver failure after liver resection in patients with Child-Pugh grade A cirrhosis. Br J Surg. 2012 Dec;99(12):1701-10. doi: 10.1002/bjs.8951. PMID 23132418
- [Derived] Li XL, Zhu XD, Xiao N, Liu XF, Xu B, Shi GM, Huang C, Shen YH, Cai JB, Zhou J, Fan J, Sun HC. A prospective study of the effect of terlipressin on portal vein pressure and clinical outcomes after hepatectomy: A pilot study. Surgery. 2020 Jun;167(6):926-932. doi: 10.1016/j.surg.2020.01.013. Epub 2020 Feb 26. PMID 32113581